CLINICAL TRIAL: NCT04748471
Title: A Phase II Trial Assessing Immunogenicity and Safety of SARS-CoV-2 Vaccine mRNA-1273 in Volunteers Aged of 65 Years or More Compared to Participants 18-45 Years Old
Brief Title: Immunogenecity and Safety of VaccinemRNA-1273 in Elderly Volunteers (Over 65 y) Compared to Younger Ones (18-45y)
Acronym: CoviCompareM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP201504; 2020-005889-34 (EudraCT Number)
Record Dates: First submitted 2021-01-24; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Prevention of COVID19
Keywords: Vaccinology; Infectiology; Vaccine; COVID-19; Immunity; Immune; Cells; Mucosal immunity; Autoimmunity
MeSH Terms: conditions — COVID-19; Autoimmune Diseases | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 18-45 years old (Experimental): 18 - 45 years old (60 volunteers), 2 injections of mRNA-1273, at day 1 and day 29
  Interventions: Biological: mRNA-1273
- 65-74 years old (Experimental): 65 - 74 years old (60 volunteers), 2 injections of mRNA-1273, at day 1 and day 29
  Interventions: Biological: mRNA-1273
- At least 75 years old (Experimental): At least 75 years old (60 volunteers), 2 injections of mRNA-1273, at day 1 and day 29
  Interventions: Biological: mRNA-1273

INTERVENTIONS:
Biological: mRNA-1273 — SARS-CoV-2 vaccine

SUMMARY:
This study aims to evaluate the immunogenicity of Moderna mRNA-1273 vaccine in volunteers aged 65 years or more compared to volunteers aged 18-45 years, over 24 months duration. It will provide necessary data on the early immunological response to the vaccine and its evolution in quantitative and qualitative terms. This study will allow establishing how aging influences the response to the vaccine and help to adapt the vaccinal plan. For instance it will suggest the necessity of a vaccination booster.

DETAILED DESCRIPTION:
Phase II, comparative, non-randomized trial assessing the immunogenicity and safety of vaccine candidate Moderna-1273 against SARS-CoV-2. A total of 180 volunteers will be included and vaccinated (2 doses, at day 1 and day 29), divided in 3 groups (60 volunteers 18 - 45 years old, 60 volunteers 65 - 74 years old, 60 volunteers at least 75 years old). Vaccinated volunteers of the three arms will be immune-monitored during 24 months via a battery of in vitro and ex vivo tests to comprehensively assess the course of humoral, cellular and mucosal immunity over time.

ELIGIBILITY:
Inclusion Criteria:

1. At least 65 years old, at least 75 years old or 18 to 45 years old, depending on the group of inclusion.
2. Healthy adults, or stable medical condition for adults with pre-existing medical conditions. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during 3 months before enrolment, nor expected to require any significant change in therapy or hospitalization for worsening disease in foreseeable future.
3. Understands and agrees to comply with the study procedures (visits, phone calls) and provides written free informed consent.
4. Able to comply with study procedures based on Investigator judgement.
5. Affiliated to a social security system, (except state medical aid)

Exclusion criteria:

1. Subject is ill or febrile (body temperature ≥ 38.0°C) within 72 prior hours or and/or symptoms suggestive of COVID-19 within the past 14 days at enrolment visit.

   (Ill or febrile participants may be re-scheduled within the inclusion period when no longer presenting symptoms)
2. History of documented COVID-19 (PCR+, antigenic test+ or chest TDM+ or serology SARS-CoV-2+) prior to first vaccine administration
3. Subjects with positive serology to SARS-CoV-2 at the enrolment visit
4. Subjects who already received another anti-SARS-CoV-2-vaccine
5. Subjects who received BCG given within the last year.
6. An immediate family member or household member of study staff.
7. Use of immunosuppressive drugs like e.g. corticosteroids at a dosage > 10mg/day (excluding topical preparations and inhalers) within 3 months prior to enrolment or 6 months for chemotherapies
8. Received immunoglobulin or other blood product within 3 months prior to enrolment or planned receipt of immunoglobulin or a blood product through study completion.
9. Received any vaccination within 4 weeks prior to first injection or plan to receive a licensed vaccine 4 weeks after the last injection.
10. History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as rush, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of allergic reaction likely to be exacerbated by any component of the anti-SARS-CoV-2-vaccine.
11. History of severe allergic event
12. Participation in another investigational clinical study (Jardé 1 or Jardé 2) within 4 weeks before the enrolment visits or planned before the study completion.
13. Known HIV, active HCV or HBV infection
14. Any pathological condition, such as cancer, which may be susceptible of reducing immunity response
15. Any bleeding disorder considered as contraindication to intramuscular injection or phlebotomy
16. The use of investigational Ig, investigational monoclonal antibodies or convalescent serum are not allowed during the study
17. Any condition which in the opinion of the investigator may interfere with the aim of the study
18. Pregnant or breastfeeding or positive pregnancy urine test at enrolment visit.
19. Woman in childbearing without efficacious contraception (in the opinion of the investigator) for 31 days after treatment (2nd vaccine injection)
20. People under legal protection measure (tutorship, curatorship or safeguard measures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-02-10 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2023-01-25 (Estimated)

PRIMARY OUTCOMES:
Titers of anti-SARS-CoV-2 Spike IgG Immunoglobulin in sera | Day 57 (28 days after second injection of mRNA-1273)
  Anti-SARS-CoV-2 Spike specific IgG Immunity acquisition

SECONDARY OUTCOMES:
Anti SARS-CoV -2 IgG, IgA and IgM (total and subclasses IgG1-4) as measured by ELISA. | From Day 1 to Month 24
  Assessment of humoral immunity-systemic response
Anti-SARS-CoV-2 neutralizing antibody (in vitro neutralisation assay. | From Day 1 to Month 24
  Assessment of humoral immunity-systemic response
Anti-SARS-CoV-2 -specific neutralizing antibody (Pseudo neutralisation assay using lentiviral phenotypes carrying specific SARS-Cov-2 proteins. | From Day 1 to Month 24
  Assessment of humoral immunity-systemic response
Fluorospot assays (TH1, TH2, TH17, Cytotoxicity). Phenotyping of antigen specific T-Cells via Mass cytometry, B cell repertoire and memory | From Day 1 to Month 24
  Assessment of cellular immunity acquisition
Mucosal SARS-CoV-2 -specific antibody via measure of sIgA, sIgM and IgG in saliva by specific home-made and commercially available ELISA assays. | From Day 1 to Month 24
  Assessment of mucosal immunity
Functionality of mucosal sIgA and sIgM by Antibody Dependent Cellular Cytotoxicity (ADCC) assay specific for SARS-CoV-2 mucosal IgA and IgM | From Day 1 to Month 24
  Assessment of mucosal immunity
Local and systemic reactogenicity | From Day 1 to Month 24
  Clinical safety evaluation
Determination of autoimmunity markers such as antibodies Anti-nuclear (unit measure: titers) | From Day 1 to Month 24
  Biological safety evaluation
Determination of autoimmunity markers such as antibodies Anti-ACL, Anti-β2-GP1, Rheumatoid factor (unit measure: U/L) | From Day 1 to Month 24
  Biological safety evaluation
Determination of autoimmunity markers such as antibodies Anti-GM1, Anti-MAG ( unit measure: pos/ne) | From Day 1 to Month 24
  Biological safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.